CLINICAL TRIAL: NCT03212612
Title: Galectin-3 in Patients With Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Magdy Mohammed, galectin-3 in women with endometriosis, Assiut University
Other Study IDs: 17100222
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Endometriosis
Keywords: Galectin-3 ,endometrosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Endometrial samples(1-2 gram) will be separated from each women during proliferative phase(days 5-15) and washed several times with 0.9% sterile saline solution to remove any blood from the tissues. The tissue samples will homogenized by tissue homogenizer at 40,000rpm. The supernatant extracts will be collected in Ependorf tubes and frozen at -80°C till analysis by ELISA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2 groups , control and cases: Groupe 1: (cases) 45 women who were found to have surgically and histolopathologically -confirmed endometriosis. Endometrial samples(1-2 gram) will be taken by laparoscopy which is the gold standard for definitive diagnosis of endometriosis.
  Group2:(control) 45women who were free of endometriosis. Endometrial samples(1-2 gram) will be taken by punch biopsy.
  Interventions: Diagnostic Test: samples obtained by laparoscopy or punch biopsy for analysis by ELISA

INTERVENTIONS:
Diagnostic Test: samples obtained by laparoscopy or punch biopsy for analysis by ELISA — Endometrial samples(1-2 gram) will be separated from each women during proliferative phase(days 5-15) by laparoscopy or punch biopsy and washed several times with 0.9% sterile saline solution to remove any blood from the tissues. The tissue samples will homogenized by tissue homogenizer at 40,000rpm. The supernatant extracts will be collected in Ependorf tubes and frozen at -80°C till analysis by ELISA

SUMMARY:
The exact cause of endometriosis is unknown ,so our study is to investigate the relationship between Galectin-3 and endometriosis by comparing between its level in healthy and endometriosis women. Also, we will measure the level of oxidative stress markers in endometrium of both healthy and endometriosis women and investigate the correlaton between them and galectin-in endometriosis women.

DETAILED DESCRIPTION:
Endometriosis is a benign gynaecological disorder with malignant biological characteristics and is defined by the presence of endometrial glands and stroma outside the uterine cavity. Ectopic endometrial cells can spread to pelvic organs such as rectum, bladder, and ovaries. The pathophysiology of endometriosis is likely to be multifactorial and to involve an interplay between several factors. (Fauser BC, Diedrich K, Bouchard P, Domínguez F, Matzuk M, 2011)

The endometrial cycle and implantation are complex processes. Alterations in levels of some regulatory molecules on the cell surface occur during the cycle tightly controlled proliferation and differentiation. Most of these regulatory molecules and mechanisms have not yet been investigated, However, Galectins , a sub family of lectins are delineated to regulate vital cell functions. (Leffler H. et al Introduction to galectins. Glycoconj j,2004) It has been shown that Gal-3 is expressed in many cell types, including endometrial cells and trophoblast cells (Riss D, Naude S 2003) . Previous studies have reported that Gal-3 is specifically expressed in endometrial cells in the secretory phase, in placental tissue during early pregnancy, and in decidua surrounding the site of implantation. Another study verified that Gal-3 plays an important role in the process of embryonic implantation (Liu YK, Hum Reprod.2009). Intracellular Gal-3 promoted proliferation and adhesion in endometrial cells(Yang H, TaylorHS,2011) .

Female reproductive system is vulnerable to the harmful effects of reactive oxygen species (ROS) that damage proteins, lipids, and DNA structure. Oxidative stress is a key factor for progression of endometriosis. Many theories have been elaborated so far to clarify endometriosis pathogenesis and oxidative stress, a result of increased production of free radicals or depletion of the body's endogenous antioxidant defense, has been implicated in its pathogenesis.

Our study is a case-control study that will be made in woman health hospital and medical biochemistry department -assiut university. We will estimate the tissue level of galectin-3 in endometrium of both healthy and endometriosis women and detect wether galectin-3 leads to or protect against endometriosis. Also, we will measure the level of oxidative stress markers in endometrium of both healthy and endometriosis women and investigate the correlaton between them and galectin-in endometriosis women.

The sample size is calculated by Epi Info 2000 software computer program. Based on the expected proportion of Galectin-3 deficiency among controls will be 20% and its increase in cases by four folds (Odd Ratio = 4) with 80% power and a confidence level 95%, the calculated sample size is 45cases and 45 controls (totally 90 women).

The data collected will include age, parity, menstrual history , present history (including symptoms of pain, bleeding and infertility), drug history , history of previous diseases and any investigations were done. The aim of the study will be explained to each participant before filling study sheet. A written consent will be obtained from those who welcome to participate in the study, then women will be divided into 2 groups.

Group1:

45women who were found to have surgically and histolopathologically -confirmed endometriosis. Endometrial samples(1-2 gram) will be taken by laparoscopy which is the gold standard for definitive diagnosis of endometriosis.

Group2:

45 women free of endometriosis. These women had normal menstrual cycles and had not received hormonal therapy within 3 months prior to sampling. Endometrial samples(1-2 gram) will be taken from them through Punch biopsy after IUD insertion.

Galectin-3 will be estimated by ELISA kit. Endometrial samples(1-2 gram) will be separated from each women during proliferative phase(days 5-15) and washed several times with 0.9% sterile saline solution to remove any blood from the tissues. The tissue samples will homogenized by tissue homogenizer at 40,000rpm. The supernatant extracts will be collected in Ependorf tubes and frozen at -80°C till analysis by ELISA.

The tissue levels of NO and TBARS (oxidative stress markers) were determined by chemical methods according to the methods descriped by Van Bezooijen et al, (1998), and Buege and Aust (1978) respectively. Also the tissue levels of catalase (CAT), glutathione (GSH) and superoxide dismutase (SOD) activity (anti oxidants) were determined by chemical methods according to the methods descriped by Clairborne ( 1985), Beutler et al. (1963) and Marklund (1985).

ELIGIBILITY:
Inclusion Criteria:

Age:20-35 years In women with endometriosis

Exclusion Criteria:

Women who have irregular menstrual cycles

Women who are pregnant, have pelvic inflammatory disease, cervical erosion, vaginal infection or coagulopathies.

Women who have liver disease, renal disease or cardiac disease that can affect level of Galectin-3.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include women aged from 20 to 35 years old in woman health hospital.
  The aim of the study will be explained to each participant before filling study sheet. A written consent will be obtained from those who welcome to participate in the study .The data collected will include age, parity, menstrual history , present history (including symptoms of pain, bleeding and infertility), drug history , history of previous diseases and any investigations were done. Then women will be divided into 2 groups, (group of cases and a control group)
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
To measure the level of Galectin-3 proteins in patients of endometriois and investigate the relationship between Galectin-3 and endometriosis by comparing between its level in healthy and endometriosis women. | 6 months
  galectin-3 level will be estimated in both healthy and endometriosis women by ELISA to iinvestigate the role of galectin-3 in etiology of endometriosis

CONTACTS AND LOCATIONS:
Overall Officials: heba magdy mohammed, Principal Investigator — faculty of medicine -aasiut university
Locations (3):
- Egypt (3):
  - Faculty of Medicine - Assiut University, Asyut
  - Faculty of Medicine -Assiut University, Asyut
  - Faculty of Medicine- Assiut University, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yang H, Yin J, Ficarrotta K, Hsu SH, Zhang W, Cheng C. Aberrant expression and hormonal regulation of Galectin-3 in endometriosis women with infertility. J Endocrinol Invest. 2016 Jul;39(7):785-91. doi: 10.1007/s40618-016-0435-7. Epub 2016 Feb 17. PMID 26886939